CLINICAL TRIAL: NCT03592134
Title: Choice and Optimal Settings of Non Invasive Respiratory Support in Preterm Newborns < 30 Gestational Weeks
Brief Title: Optimal Settings of Non Invasive Respiratory Support in Preterm Newborns
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hôpital Necker-Enfants Malades (Other)
Responsible Party: Principal Investigator, Brigitte Fauroux, Professor, Hôpital Necker-Enfants Malades
Other Study IDs: 2017-A00535-48
Record Dates: First submitted 2018-07-05; First posted 2018-07-19 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Preterm Infant; Respiratory Distress Syndrome
MeSH Terms: conditions — Premature Birth; Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Clinical settings: Infants with the choice of the non respiratory support and settings of the non respiratory support defined by clinical practice (nocturnal gas exchange, apneas, bradycardia, oxygen desaturation)
- Physiological settings: Infants with the choice of the non respiratory support and settings of the non respiratory support defined by the measurement of work of breathing
  Interventions: Other: esophageal pressure measurement

INTERVENTIONS:
Other: esophageal pressure measurement — Measurement of esophageal pressure to determine the optimal non invasive respiratory support
  Groups: Physiological settings

SUMMARY:
Noninvasive respiratory supports (NRS), such as continuous positive airway pressure (CPAP), noninvasive ventilation, high flow nasal cannula (HFNC) or nasal oxygen (O2), are commonly used in preterm newborns hospitalized in neonatal intensive care unit. However, given the lack of validated criteria, clinicians usually choose the NRS according to clinical parameters and patients' comfort. Several studies have demonstrated the interest of the measurement of the work of breathing (WOB) to optimize the settings of NRS in children, but no study has already demonstrated the utility of WOB to optimize the settings of NRS in preterm infants. Therefore, the aim of this study is to measure the WOB during the utilisation of three different NRS (CPAP, HFNC, O2), in order to optimize the choice of the type and settings of NRS in a randomized group of 30 newborns born prematurely before 30 gestational weeks and still requiring NRS at 29 post conceptual weeks. Moreover, the investigators will compare in the newborns with the optimized NRS by WOB vs. a standard care control group (NRS type and settings determined as clinical routine): 1) the respiratory morbidity and mortality one month after the initial assessment, and at the time of hospital discharge (or transfer) or at 36 weeks of age corrected (whatever comes first), 2) the weaning time of the NRS, 3) the incidence and severity of broncho-pulmonary dysplasia (BPD) at 36 weeks of age corrected. Indeed, incidence of BPD is still around 40% in premature infants born before 28 gestational weeks. The hypothesis of the investigators' study is that the optimization of the type and settings of the NRS could reduce the weaning delay and contribute to reduce the incidence and severity of BPD in premature newborns.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants born between 23 and 30 GA
* Aged over 29 weeks of corrected age at the time of assessment and needing a non invasive respiratory support since at least 4 weeks of age

Exclusion Criteria:

* Hemodynamic and/or neurologic instability
* Invasive ventilation
* Congenital cardiopathy and/or significant patent ductus arteriosus
* Sedation
* Congenital pulmonary disease and/or other malformations

Ages: 4 Weeks to 6 Weeks | Sex: All
Age Groups: Child
Study Population: Preterm infants needing a non invasive respiratory support after 4 weeks of life
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-02-22 (Actual); Primary Completion 2018-09-21 (Estimated); Study Completion 2018-11-09 (Estimated)

PRIMARY OUTCOMES:
Maximal variation of esophageal pressure | at participant inclusion day 1
  Maximal variation of esophageal pressure will be compared for the different respiratory supports and the different settings

SECONDARY OUTCOMES:
occurrence of bronchopulmonary dysplasia at 36 Gestational age (GA) | From 2 to 7 weeks after participant's inclusion (day 1)
need for nutritional support | From 2 to 7 weeks after participant's inclusion (day 1)
definitive weaning delay | From 2 to 7 weeks after participant's inclusion (day 1)
  weaning from noninvasive respiratory support and oxygen supplementation

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte Fauroux, MD, PhD, Principal Investigator — AP-HP Hopital Necker
Locations (1):
- AP-HP Hopital Necker, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Liptsen E, Aghai ZH, Pyon KH, Saslow JG, Nakhla T, Long J, Steele AM, Habib RH, Courtney SE. Work of breathing during nasal continuous positive airway pressure in preterm infants: a comparison of bubble vs variable-flow devices. J Perinatol. 2005 Jul;25(7):453-8. doi: 10.1038/sj.jp.7211325. PMID 15858606
- [Result] Shetty S, Hickey A, Rafferty GF, Peacock JL, Greenough A. Work of breathing during CPAP and heated humidified high-flow nasal cannula. Arch Dis Child Fetal Neonatal Ed. 2016 Sep;101(5):F404-7. doi: 10.1136/archdischild-2015-309310. Epub 2016 Jan 14. PMID 26769758
- [Result] de Jongh BE, Locke R, Mackley A, Emberger J, Bostick D, Stefano J, Rodriguez E, Shaffer TH. Work of breathing indices in infants with respiratory insufficiency receiving high-flow nasal cannula and nasal continuous positive airway pressure. J Perinatol. 2014 Jan;34(1):27-32. doi: 10.1038/jp.2013.120. Epub 2013 Sep 26. PMID 24071905
- [Result] Saslow JG, Aghai ZH, Nakhla TA, Hart JJ, Lawrysh R, Stahl GE, Pyon KH. Work of breathing using high-flow nasal cannula in preterm infants. J Perinatol. 2006 Aug;26(8):476-80. doi: 10.1038/sj.jp.7211530. Epub 2006 May 11. PMID 16688202